CLINICAL TRIAL: NCT05294081
Title: EFFECT-BACK: Tackling Back Pain - Effects of Exposure Therapy and Cognitive Behavioural Therapy for Chronic Back Pain
Brief Title: EFFects of EXPosure and Cognitive-behavioural Therapy for Chronic BACK Pain
Acronym: EFFECT-BACK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kaiserslautern-Landau (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFECT-BACK1/2022
Record Dates: First submitted 2022-03-02; First posted 2022-03-24 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Cognitive Behavioural Therapy; Exposure; Fear Avoidance; Cognitive Behavioural Therapy in chronic low back pain; Exposure in vivo in chronic low back pain
MeSH Terms: interventions — Implosive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicentre, randomised, controlled, open-label, two-arm intervention study with a parallel group design.
  Two parallel groups are formed, the intervention group receives 10 sessions of EXP therapy, the control group receives 10 sessions of CBT.
  The assignment to the therapy methods is randomised. This is a multicentre study, the study will be conducted at 5 centres throughout Germany. A total of 380 patients will be included. Per study arm, 190 patients must be included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (EXP) (Experimental): Exposure in vivo for fear avoidant chronic low back pain patients. This treatment means that the individual is exposed to movements and tasks that have been avoided due to fear of (re)injury. The treatment begins after three educational lessons including the rational and developing a fear hierarchy. Exposure phase includes 10 exposures sessions which are highly individualized. Behavioral experiments can be included to correct catastrophic misinterpretations. The main purpose of this intervention type is to reduce pain related disability via diminishing fear avoidance.
  Interventions: Behavioral: Exposure therapy
- Cognitive Behavioural Therapy (CBT) (Active Comparator): Cognitive behavioural psychotherapy for fear avoidant chronic low back patients. The therapy is modularized in three main parts. The educational lesson is followed by the module graded activity which represents the behavioral part of the program. The second module comprises relaxation. And the last part contains cognitive interventions. Cognitive behavioural intervention techniques are employed to support the patient in the process of coping with chronic pain: i.e. reduction of disability and improving functional ability.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Exposure therapy — 10 sessions based on an individualized pain hierarchy
  Arms: Exposure (EXP)
Behavioral: Cognitive behavioral therapy — 10 sessions with graded activity, relaxations techniques and cognitive interventions
  Arms: Cognitive Behavioural Therapy (CBT)

SUMMARY:
The overall aim of the present study is to compare two different psychological methods, Cognitive Behavioural Therapy (CBT) and Graduated Exposure in vivo (EXP) in the treatment of chronic back pain with regard to effectiveness and improvement of pain related disability.

Exploratory research will also be conducted to identify predictors of which patient groups benefit more from which method. This should optimise treatment options and create effective treatment offers for subgroups of pain patients.

Exposure therapy is an effective and economical treatment modality and was shown in a previous pilot study to be superior to CBT in reducing perceived movement limitation. CBT, on the other hand, appeared to be more effective in establishing coping strategies. With the help of the current study it should be possible to compare the effectiveness of both treatment methods and, in perspective, to identify those patient groups that benefit from exposure therapy and thus create a tailor-made treatment programme for subgroups of pain patients.

A total of 380 patients (age: ≥ 18) with chronic back pain and a sufficient degree of impairment will be included and analysed in the study.

DETAILED DESCRIPTION:
According to a recently published study by the Robert Koch Institute with over 62 000 participants, one in six men (17.1%) and one in four women (24.4%) in Germany reported having suffered from chronic low back pain (CLBP) in the last 12 months. CLBP is a major cause of medical costs, absenteeism and disability. Despite apparent advances in medical care, the prevalence of CLBP continues to rise.

According to current guidelines, most of the commonly offered treatments such as injections or surgery are ineffective; only pharmacotherapy shows small effects but carries a high risk of side effects.

Cognitive behavioural therapy (CBT), multidisciplinary approaches with psychological treatment components such as CBT and exercise, supported by psychological elements, improve pain and condition-related disability in the long term. Disappointingly, however, in most studies the effects of multidisciplinary or psychological treatment approaches are small to moderate, and in the case of multidisciplinary approaches, do not always justify the high costs of inpatient programmes. In outpatient care, specific psychological services in addition to pharmacotherapy and physiotherapy are rare.

EXP treatment for pain is a rarely used psychological treatment that specifically addresses the avoidance of physical activity in people with CLBP. In a previous pilot study with 88 participants, the investigators conducted for the first time a short (10 sessions) and a longer (15 sessions) outpatient EXP therapy programme and compared it with a standard 15-session CBT programme:

* EXP was more effective than CBT in reducing movement-related impairment.
* EXP-short outperformed EXP-long in efficiency after 10 sessions, meaning that individuals improved faster when offered fewer sessions.
* EXP could be safely delivered in the outpatient psychological setting, however CBT was more effective than EXP in improving coping strategies.

A specific behavioural measure, the "BAT-BACK" test, successfully identified participants who benefited from EXP in terms of a reduction in pain-related impairment. Therefore, in the future, EXP therapy could be a tailored treatment option to achieve better treatment outcomes in subgroups of CLBP patients. However, studies with more participants are needed to further clarify whether EXP is successful and for which subgroup of patients. The proposed study would be the first to aim to find out which patient group is more likely to benefit from EXP and which from CBT.

Research question and rationale for the project:

Society is currently faced with the challenge of a widespread disease without being able to offer satisfactory treatment options. A comparison of an already established treatment method (CBT) with a still less known and used treatment method (EXP) should create starting points here. In addition, tailoring chronic pain treatment specifically to subgroups of pain patients could improve care.

In addition, EXP therapy is a promising and cost-effective treatment option that could easily be incorporated into multidisciplinary programmes for inpatients or offered by outpatient psychotherapists as part of the newly established 12-hour brief psychotherapy. In order to validate the preliminary results of the pilot study and to answer open questions, a multicentre study with a larger number of participants is implemented.

The study should also lead to a larger number of therapists trained in EXP therapy in different regions in Germany and to an increase in the visibility of the treatment manuals and could lead to a more frequent use of EXP for the benefit of the CLBP population. By publishing the results, the investigators hope to raise awareness, especially among psychological psychotherapists, that brief, manualised, focused treatments may be sufficient to reduce the burden of chronic pain. The identification of predictors will help all practitioners involved in the treatment of chronic pain to identify those patients who are more likely to benefit from EXP and those who are more likely to benefit from CBT.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (duration > 6 months, pain on most days of the week)
* Sufficient level of disability, as defined by QBPDS ≥ 15 (Quebec Back Pain Disability Scale)
* Age 18 and above
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* Back surgeries during the last six months or planned surgeries
* Red Flags
* inability to read or write in German
* pregnancy
* severe alcohol or drug addiction
* psychotic disorders
* another current psychological treatment
* physical inability to attend sessions
* parallel participation in another intervention study

Depression will be controlled for, medication will be required to stay stable until Follow-up and any changes will be controlled for, on-demand ("rescue") medication will be not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain related disability | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months after Posttest and 2 years after Posttest)
  Clinically significant change in pain-related impairment at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Quebec Back Pain Disability Scale (QBPDS). Each item is scored from 0 to 5 (0 = not difficult at all, 5 = unable to do). Higher total scores reflect higher disability.

SECONDARY OUTCOMES:
Change in pain disability | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Clinically significant change in pain-related impairment at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Pain Disability Index (PDI). Each item is scored from 0 to 10 (0 = no disability, 10 = maximum disability). Higher total scores reflect higher interference of pain with daily activities.
Change in pain intensity | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Clinically significant change in pain intensity at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  adjusted 11-point Scale of the German Pain Questionaire (Deutscher Schmerzfragebogen, DSF). 3 Items, each item is scored from 0 to 10 (e.g. 0 = no pain, 10 = strongest pain). A higher score reflects stronger pain.
Change in coping | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in coping at the end of therapy and at 6-month and 2-years follow-up compared to baseline.
  Coping scale from the German questionnaire for the assessment of pain processing (Fragebogen zur Erfassung der Schmerzverarbeitung, FESV-BW). Each item is scored from 1 to 6 (1 = not true at all, 6 = completely true). Higher total scores reflect more frequent use of different coping strategies.
Change in emotional distress | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in depression at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Depression scale of the Hospital Anxiety and Depression Scale (HADS). Each item is scored from 0 to 3. Higher total scores reflect stronger anxiety or depressiveness.
Change in pain catastrophizing | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in catastrophizing at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Pain Catastrophizing Scale (PCS). Each item is scored on a scale of 0 to 4 (0 = not at all, 4 = all the time). Higher total scores reflect more catastrophising thoughts.
Change in kinesiophobia | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in kinesiophobia at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Photo Series of Daily Activities (PHODA). Each item is scored from 0 to 100 (0 = not harmful at all, 100 = extremely harmful). Higher scores reflect higher perceived harmfulness.
Change in pain anxiety | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in pain anxiety avoidance at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Pain Anxiety Symptom Scale (PASS-20). Each item is scored from 0 to 5 (0 = never, 5 = always). Higher total scores reflect more fear of pain.
Change in psychological inflexibility | from Baseline to Posttest (an expected average of 15 weeks) to Follow Up Assessments (an expected average of 6 months and 2 years after Posttest)
  Change in psychological inflexibility at the end of therapy and at 6-months and 2-years follow-up compared to baseline.
  Psychological Inflexibility in Pain Scale (PIPS). Each item is scored from 1 to 7 (1 = never true, 7 = always true). Higher total scores reflect higher inflexibility because of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Glombiewski, Prof. Dr., Study Director — RPTU Kaiserslautern - Landau, Department of Clinical Psychology and Psychotherapy
Locations (5):
- Germany (5):
  - RPTU Kaiserslautern- Landau, Landau, RLP
  - Essener Rückenschmerzzentrum, Universitätsklinikum Essen, Essen
  - Schmerzzentrum, Ruprechts - Karls Universität Heidelberg, Heidelberg
  - Poliklinische Institutsambulanz für Psychotherapie, Mainz
  - Phillips-Universität Marburg, Marburg

REFERENCES:
- [Background] Kuntz B, Hoebel J, Fuchs J, Neuhauser H, Lampert T. [Social inequalities in the prevalence of chronic back pain among adults in Germany]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2017 Jul;60(7):783-791. doi: 10.1007/s00103-017-2568-z. German. PMID 28516263
- [Background] van Tulder M, Koes B. Chronic low back pain. Am Fam Physician. 2006 Nov 1;74(9):1577-9. No abstract available. PMID 17111899
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Bernstein IA, Malik Q, Carville S, Ward S. Low back pain and sciatica: summary of NICE guidance. BMJ. 2017 Jan 6;356:i6748. doi: 10.1136/bmj.i6748. No abstract available. PMID 28062522
- [Background] Eccleston C, Morley SJ, Williams AC. Psychological approaches to chronic pain management: evidence and challenges. Br J Anaesth. 2013 Jul;111(1):59-63. doi: 10.1093/bja/aet207. PMID 23794646
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain. Cochrane Database Syst Rev. 2014 Sep 2;2014(9):CD000963. doi: 10.1002/14651858.CD000963.pub3. PMID 25180773
- [Background] Glombiewski JA, Holzapfel S, Riecke J, Vlaeyen JWS, de Jong J, Lemmer G, Rief W. Exposure and CBT for chronic back pain: An RCT on differential efficacy and optimal length of treatment. J Consult Clin Psychol. 2018 Jun;86(6):533-545. doi: 10.1037/ccp0000298. PMID 29781651
- [Background] Holzapfel S, Schemer L, Riecke J, Glombiewski JA. Behavioral Test (BAT-Back): Preliminary Evidence for a Successful Predictor of Treatment Outcome After Exposure Treatment for Chronic Low Back Pain. Clin J Pain. 2021 Apr 1;37(4):265-269. doi: 10.1097/AJP.0000000000000920. PMID 33555697
- [Background] Hasenbring MI, Verbunt JA. Fear-avoidance and endurance-related responses to pain: new models of behavior and their consequences for clinical practice. Clin J Pain. 2010 Nov-Dec;26(9):747-53. doi: 10.1097/AJP.0b013e3181e104f2. PMID 20664333
- [Background] de Jong JR, Vlaeyen JWS, Onghena P, Cuypers C, den Hollander M, Ruijgrok J. Reduction of pain-related fear in complex regional pain syndrome type I: the application of graded exposure in vivo. Pain. 2005 Aug;116(3):264-275. doi: 10.1016/j.pain.2005.04.019. PMID 15964686
- [Derived] Vogt R, Haas J, Baumann L, Sander A, Klose C, Riecke J, Rief W, Bingel U, Maser D, Witthoft M, Kessler J, Zugaj MR, Ditzen B, Glombiewski JA. EFFects of Exposure and Cognitive behavioral Therapy for chronic BACK pain ("EFFECT-BACK"): study protocol for a randomized controlled trial. Trials. 2024 Mar 11;25(1):176. doi: 10.1186/s13063-024-08017-9. PMID 38468293

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Main project (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT05294081/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Amendment (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT05294081/Prot_SAP_001.pdf